CLINICAL TRIAL: NCT00157235
Title: A Randomized, Double Blind , Placebo Controlled Trial to Compare the Effect of Tiotropium Inhalation Capsules on Exercise Tolerance in Patients With COPD Participating in 8 Weeks of Pulmonary Rehabilitation
Brief Title: Effect of Tiotropium Inhalation Capsules (Spiriva) on Exercise Tolerance in COPD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.247
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: Tiotropium bromide

SUMMARY:
The objective of this trial is to determine whether tiotropium inhalation capsules (Spiriva, Bromuro de Tiotropio), compared to placebo, enhances the improvement in exercise tolerance seen in patients with chronic obstructive pulmonary disease (COPD) who participate in pulmonary rehabilitation.

DETAILED DESCRIPTION:
This is an 25-week multicenter, single country, randomised, double-blind, placebo-controlled, parallel group study to compare the efficacy of tiotropium inhalation capsules (Spiriva, Bromuro de Tiotropio) in patients with COPD participating in a pulmonary rehabilitation program.

Following an initial screening, patients will perform a six minute walk test (Visit 1) and enter a 4-week run-in period. Patients will subsequently be randomized to tiotropium or placebo inhalation capsules taken once daily in the morning for the next 25 weeks. After successfully completing 4 weeks of study drug self-administration, patients will enter a period of pulmonary rehabilitation.

Pulmonary rehabilitation will include aerobic lower limb exercise 3 times weekly for 8 weeks. After the last pulmonary rehabilitation session, patients will continue on study medication for a 12 week follow-up period.

Six minute walk tests will be repeated during the run-in period at Week 0 (Visit 2) and Week 4 (Visit 3), at the conclusion of the 8 weeks of pulmonary rehabilitation (Visit 6) and the 12 weeks of follow-up (Visit 9).

Pulmonary function testing will be conducted prior to the start of therapy at Visit 1 and at Visits 2 (week 0 ), 3 (week 4 ), 6 (week 13 ) and 9 (week 25 ).

Study Hypothesis:

The null hypothesis is that there is no difference in the increase in six minute walk distance between tiotropium and placebo groups following 8 weeks pulmonary rehabilitation program. The alternative hypothesis is that tiotropium with pulmonary rehabilitation increases six minute walk distance more than placebo with pulmonary rehabilitation. However, the two-sided test of hypothesis will be performed at 0.05 level of significance.

Comparison(s):

The primary endpoint is the six minute walk distance at visit 6. This endpoint will be compared between tiotropium and placebo using an analysis of covariance model with treatment, center and baseline (six-minute walk distance measured at visit 2 prior to dosing) as a covariate. Fifty-four meters has been determined to be the difference in six minute walk distance between tiotropium (Spiriva, Bromuro de Tiotropio) and placebo at 5% level of significance with at least 80% power using a two-tailed t-test.. .

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with FEV1 less 60% of predicted FEV1 less 70% of FVC.

Exclusion Criteria:

* Patients with any respiratory infection in the six weeks prior to the Screening Visit or during the run-in period (between Visits 1 and 2).
* Patients with a recent history (i.e., 6 months - or less) of myocardial infarction.
* Patients with any cardiac arrhythmia requiring drug therapy in the past year or who have been hospitalized for heart failure within the past three years.
* Patients with symptomatic benign prostatic hypertrophy or bladder neck obstruction.
* Patients with known narrow-angle glaucoma.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234
Dates: Start 2002-09; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Change in six minute walk distance after 8 weeks of pulmonary rehabilitation. | week 13

SECONDARY OUTCOMES:
Individual FEV1 measurement | week 4, 13, 25
Individual FVC measurement | week 4, 13, 25
St. George's Hospital Respiratory Questionnaire (SGRQ) | Time Frame: week 4, 13, 25
Transition dyspnea index | week 4, 13, 25
COPD symptom scores (wheezing, shortness of breath, coughing and tightness of chest | week 4, 13, 25
Amount of salbutamol therapy used during the treatment period | 25 weeks
Number and length of exacerbations of COPD | 25 weeks
Physician's global evaluation | week 4, 13, 25
Patient peak flow rates (PEFR) twice daily | 25 weeks
Patient activity measurement | week 4, 9, 13, 17, 21, 25
Six minute walk distance | week 13, 25
Occurrence of adverse events | 25 weeks
Changes from baseline in Pulse rate and blood pressure in conjunction with spirometry | 25 weeks
Changes in the physical examination from baseline and at the conclusion of patient participation in the trial | 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — BI Italy
Locations (12):
- Italy (12):
  - Fondazione "S. Maugeri", Bari
  - Azienda Sanitaria Locale, Casorate Primo (PV)
  - Arcispedale S. Anna, Ferrara
  - U.O. dimedicina Preventiva del Lavoro, Genova
  - Fondazione Maugeri, Gussago (BS)
  - Universita degli Studi di Pisa, Pisa
  - Fondazione Don Gnocchi, Pozzolatico (FI)
  - Azienda Ospedaliera S. Camillo Forlanini, Roma
  - Fondazione S. Maugeri, Telese Terme (BN)
  - Fondazione "S. Maugeri", Tradate (VA)
  - Ospedali Riuniti di Trieste, Trieste
  - Casa di Cura San Raffaele, Velletri (Roma)

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/19281092